CLINICAL TRIAL: NCT07118046
Title: Comparison of Fluoroscopy-only vs. Electroanatomic Mapping Strategies for Pulmonary Vein Isolation With Balloon-based Pulsed-field Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Rodríguez Muñoz (Other)
Responsible Party: Sponsor-Investigator, Daniel Rodríguez Muñoz, PhD and Medical Doctor Consultant in Cardiac Electrophysiology, Principal Investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PFA Balloon -SWEET Single Shot
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: pulmonary vein isolation; atrial fibrillation; pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All events related to the dual primary efficacy outcomes and primary safety outcome will be reviewed by an independent committee. These physicians will be responsible for reviewing the acute and chronic (>30 days) left atrial maps. Their role will be to determine PVI status and to define the type of adverse event according to its severity and relevance to the study. This committee will consist of three electrophysiologists who will not participate in the ablation or remapping procedures and who will be blinded to the characteristics of the index procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoroscopy only (Active Comparator): Fluoroscopy-only guidance throughout the procedure
  Interventions: Device: Pulmonary vein isolation
- Fluoroscopy and electroanatomic mapping (Experimental): Both fluoroscopy and electroanatomic mapping guidance
  Interventions: Device: Pulmonary vein isolation

INTERVENTIONS:
Device: Pulmonary vein isolation — Pulsed field ablation for pulmonary vein isolation in atrial fibrillation ablation

SUMMARY:
We designed a study to evaluate the impact of a two systematic strategies for PVI with the octaspline, balloon-based PFA (B-PFA) catheter. We hypothesized that the addition of electroanatomic guidance is non-superior to fluoroscopy-only guidance in achieving durable PVI.

DETAILED DESCRIPTION:
Study design This is a single-center, randomized clinical study enrolling consecutive paroxysmal or persistent AF patients undergoing PVI with a B-PFA catheter (ClinicalTrials.gov identifier: pending). Patients will be randomized in a 1:1 basis to a fluoroscopy-only strategy vs. a strategy based on the same fluoroscopy workflow but with the addition of electroanatomic mapping (EAM).

Procedures will be carried out under deep sedo-analgesia with propofol and fentanyl. Patients will be scheduled for systematic, invasive remapping of the left atrium (LA) and pulmonary veins (PVs) a minimum of 30 days after index ablation, regardless of recurrence status.

The study will be carried out in University Hospital 12 de Octubre, a tertiary academic hospital, and has already received approval from the corresponding Institutional Review Board (code 23/208, mod. 2).

Patient data will be handled according to the current General Data Protection Regulation 2016/679 of the European Parliament (EU-GDPR) and the Council of 27 April 2016 on Personal Data Protection as well as national and local regulations regarding patient autonomy, and rights and obligations in terms of information and clinical documentation.

After a run-in phase of 10 cases per operator, 96 patients will be consecutively enrolled during a 4-month period (Figure 1).

Randomization Patients who meet all eligibility criteria and provide informed consent will be assigned in a 1:1 ratio to one of two treatment arms: (1) PVI using fluoroscopy-only as guidance (control group) or (2) PVI guided by fluoroscopy with the addition of EAM (experimental group). Randomization will be performed electronically at each participating center via the Research Electronic Data Capture (REDCap®) platform (Vanderbilt University, Nashville, TN, USA). A computer-generated permuted block sequence, with stratification by AF presentation (paroxysmal or persistent), will be used to ensure balanced allocation.

Study population Patients ≥18 years old, diagnosed with paroxysmal or persistent AF and clinical indication to undergo PVI will be included. Exclusion criteria are prior PVI or left atrial linear ablation, severe frailty or life expectancy <1 year, unwillingness or inability to provide informed consent, ablation at sites beyond PVI or indication for additional electrophysiological study, contraindication or intolerance to heparin, presence of left atrial thrombus, congenital heart disease, and pregnancy, ongoing or planned in the following 6 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Diagnosed with paroxysmal or persistent AF
* Clinical indication to undergo PVI

Exclusion Criteria:

* Prior PVI or left atrial linear ablation
* Severe frailty or life expectancy <1 year
* Unwillingness or inability to provide informed consent
* Ablation at sites beyond PVI or indication for additional electrophysiological study
* Contraindication or intolerance to heparin
* Presence of left atrial thrombus
* Congenital heart disease
* Pregnancy, ongoing or planned in the following 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Durable PVI (per vein) | 30 days after index procedure
  proportion of pulmonary veins durably isolated (i.e.: more than 30 days after index procedure);
Durable PVI (per patient) | 30 days after index procedure
  proportion of patients with all pulmonary veins durably isolated (i.e.: more than 30 days after index procedure);

SECONDARY OUTCOMES:
Fluoroscopy exposure | At index procedure
  fluoroscopy time during index procedure
PFA reversibility | 30 days after index procedure
  area of reversible electroporation, measured by comparison between acute (after index procedure) and chronic (>30 day after index procedure) left atrial remapping

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rodriguez, MD PhD, Principal Investigator — University Hospital 12 de Octubre
Locations (1):
- University Hospital 12 de Octubre, Madrid, Madrid, Spain